CLINICAL TRIAL: NCT05584280
Title: Systematic Post-Implementation Evaluation of Stents
Acronym: SPECS
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: SPECS - 01
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-10

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Promus stent on shelf: Control
  Interventions: Device: Promus stent on shelf
- Orsiro stent on shelf: Treatment
  Interventions: Device: Orsiro stent on shelf

INTERVENTIONS:
Device: Orsiro stent on shelf — Cluster randomization to Orsiro stent on shelf vs. control
  Groups: Orsiro stent on shelf
Device: Promus stent on shelf — Cluster randomization to Promus stent on shelf vs. treatment
  Groups: Promus stent on shelf

SUMMARY:
To conduct a quality assurance project to establish the differences in health care processes and cost effectiveness of having the thin-strut Orsiro stent versus the thicker strut Promus stent on the shelf (i.e. as the most accessible stent).

DETAILED DESCRIPTION:
Background:

Individual patient-level randomized trials have suggested that the ultrathin strut Orsiro stent is associated with a lower risk of adverse ischemic events than the thin strut Promus stent. However, there are theoretical advantages of each stent in regards to usability, delivery and radial strength.

Study design:

The SPECS trial is a prospective, open-label, cross-sectional, cluster randomized quality assurance project, in which cardiac catheterization laboratories (hereafter referred to as center) in Västra Götaland Sweden will participate. Each week each center will place either Orsiro or Promus in the shelf in the cath lab as the most accessible stent (their workhorse stent). The specific stent to be placed on the shelf at each center each week will be randomly decided.

All patients will be treated according to local treatment guidelines and at the discretion of the interventional cardiologists, including the choice of stents.

The patients will be identified via the Swedish Web-System for Enhancement and Development of Evidence-Based Care in Heart Disease Evaluated According to Recommended Therapies (SWEDEHEART) registry. The events at will be identified and extracted from Patient registry (Socialstyrelsen), Population registry (Folkbokföringen), Causes of death registry (Socialstyrelsen). Stent usage will be monitored via SWEDEHEART and local databases (stents for which the package was opened but the stent discarded).

Study population:

Patients undergoing percutaneous coronary intervention (PCI) in Västra Götaland.

Primary objectives:

To investigate the cost-effectivess of placing either thin or thick strut stents on the shelf in the cath lab.

To investigate the weekly costs associated with placing either thin or thick strut stents on the shelf in the cath lab.

All outcomes will be tracked over time to assess whether greater experience with the thin strut stents results in changes in any cost differences over time.

If a sufficient number of patients are treated over the course of the project, retrospective analyses may be conducted using the assigned shelf stent as an instrument for assessing the effect of thin vs. thick stents on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PCI at any hospital participating in the study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing PCI at any hospital participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cost effectiveness ratio (percent) | 1 year
  Cost effectiveness of Orsiro compared to Promus on shelf.

SECONDARY OUTCOMES:
How long time did the procedure take? | During the procedure
  Procedure time (continuous variable)
How many other stents were used? | During the procedure
  Proportion of other stents used (percent)
How many additional units were needed? | During the procedure
  Number of adjunct devices used
How many patients were treated? | 1 week
  Number of patients treated
Composite of all-cause death, myocardial infarction, or coronary revascularization | 1- year
  Cumulative risk of death, myocardial infarction, or coronary revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Kardiologen, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided